CLINICAL TRIAL: NCT02349308
Title: Post Marketing Surveillance of the CentrosFLO™ Tunneled IJ Catheter for Dialysis
Brief Title: Post Marketing Surveillance of the CentrosFLO™ Tunneled IJ Catheter
Acronym: MCENPS
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013224
Record Dates: First submitted 2014-09-23; First posted 2015-01-28 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Dialysis Catheter
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CentrosFLO Long Term Hemodialysis Catheter: Schedule placement of catheter. Arterial tip of the catheter should be placed at or just above the junction of the right atrium and superior vena cava, with the arterial lumen on the left side of the catheter. The venous limb will extend into the right atrium. Catheter will be locked with the usual heparin lock solution for a newly placed catheter (at least 500 units per lumen). Fluoroscopic images will document tip position.
  Interventions: Device: CentrosFLO Long Term Hemodialysis Catheter

INTERVENTIONS:
Device: CentrosFLO Long Term Hemodialysis Catheter

SUMMARY:
The purpose of this study is to demonstrate the stability of blood flow with the CentrosFLO catheter, during intermittent dialysis over a period of 6 months after placement.

DETAILED DESCRIPTION:
The CentrosFLO™ Tunneled Dialysis Catheter is a 15F dual-lumen, double-D shaped catheter similar to other "split tip" catheters in the market: outflow ("arterial") and return ("venous") lumens that separate, a subcutaneous Dacron® cuff, extension sets with clamps and caps, and construction from Carbothane® material. The CentrosFLO™ catheter contains two small pressure-relief holes near the tips.

The main difference of the CentrosFLO catheter is in the design of the tip. Current "split tip" catheters have two free ends that diverge, but are each essentially straight segments. In the CentrosFLO catheter the arterial lumen bends in an arc back towards the venous lumen, and the venous lumen bends towards the arterial lumen. As a result, the catheter has two curved surfaces that will rest against the vena cava wall to automatically "center" the catheter within the vein. The contact points of the catheter against the vena cava wall should be smaller and more disperse than with current straight-tip or split catheters. The following drawing demonstrates the design of the catheter, showing the current recommendation that the arterial port always be to the left.

The goal of the study is to demonstrate the stability of blood flow with the CentrosFLO catheter, during intermittent dialysis over a period of 6 months after placement. The investigators plan to enroll 10 patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are initiating or continuing in-center intermittent hemodialysis who are scheduled to receive a tunneled dialysis catheter in the right or left internal jugular vein
* The patients may have had a prior tunneled catheter for dialysis in the right IJ site.
* Patients will be expected to need use of the catheter for more than 45 days

Exclusion Criteria:

* Patients in whom the catheter is planned to be placed into the same site as an existing catheter, by over-the-wire catheter exchange
* Patients unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who are initiating or continuing in-center intermittent hemodialysis who are scheduled to receive a tunneled dialysis catheter in the right or left internal jugular vein. The patients may have had a prior tunneled catheter for dialysis in the right IJ site.Patients will be expected to need use of the catheter for more than 45 days
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Stability of hydraulic resistance measured as normalized arterial pressure in mmHg/mL/min by dialysis flow meter weekly for up to six months | 1.5 years
  Stability of hydraulic resistance measured as normalized arterial pressure in mmHg/mL/min by dialysis flow meter weekly for up to six months

SECONDARY OUTCOMES:
Secondary Endpoint: Incidence of patency failure defined as blood flow rate below 300 mL/min or removal of catheter for failure of flow at any time during the study. | 1.5 years
  Incidence of patency failure defined as blood flow rate below 300 mL/min or removal of catheter for failure of flow at any time during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ash, Principal Investigator — Consulting Physican
Locations (7):
- United States (7):
  - Angiocare, Tucson, Arizona
  - Arrowhead Regional Medical Center, Colton, California
  - Olive View- UCLA Medical Center, Los Angeles, California
  - IU School of Medicine, Indianapolis, Indiana
  - IU Health Arnett, Lafayette, Indiana
  - Sierra Nephrology, Reno, Nevada
  - OSU Medical Center, Columbus, Ohio